CLINICAL TRIAL: NCT00247728
Title: A Randomized, Multi-centre, Efficacy Evaluation of PI-88 in Patients With Hepatocellular Carcinoma After Hepatectomy - A Phase II Study
Brief Title: PI-88 in Hepatocellular Carcinoma After Hepatectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cellxpert Biotechnology Corp. (Industry)
Collaborators: Medigen Biotechnology Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MG 002; PR88204 (Other: Alternate protocol identifier set by company)
Record Dates: First submitted 2005-11-01; First posted 2005-11-02 (Estimated); Results first posted 2020-11-12 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Carcinoma, Hepatocellular
Keywords: PI-88; post resection hepatoma; adjuvant therapy; hepatectomy; hepatoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — phosphomannopentaose sulfate

ARMS (3):
- Untreated Control (No Intervention): Untreated control arm
- 160 mg PI-88/Day (Experimental): PI-88 160 mg/day SC injection
  Interventions: Drug: PI-88
- 250 mg PI-88/Day (Experimental): PI-88 250 mg/day SC injection
  Interventions: Drug: PI-88

INTERVENTIONS:
Drug: PI-88 — Once-daily SC injection for four consecutive days per week, for 3 weeks out of every 4 weeks
  Arms: 160 mg PI-88/Day; 250 mg PI-88/Day

SUMMARY:
The purpose of this study is to evaluate the efficacy of PI-88 to inhibit or reduce tumor recurrence in patients with hepatocellular carcinoma following hepatectomy.

DETAILED DESCRIPTION:
Although early diagnosis and treatment improve survival, hepatocellular carcinoma (HCC) is rarely cured and recurs frequently after regional therapy or transplantation. Hepatic resection can improve 5-year recurrence-free survival by up to 25%. Micrometastases of HCC have been detected by molecular techniques in 88% of patients at the time of surgery, and probably cause postoperative recurrence. Efforts to reduce the risk of recurrence after a curative resection have been tried, including various regimens of adjuvant and neoadjuvant therapy.

In this study , an anti-angiogenic agent, PI-88, is being used as an adjuvant therapy for HCC patients after curative hepatic resection. The efficacy endpoints, including tumour non-recurrence rate, time to first recurrence and 1-year survival rate are being evaluated. Several risk factors associated with tumour recurrence are also being analysed.

ELIGIBILITY:
Inclusion Criteria:

* Patients have voluntarily given written informed consent
* Age ≥ 18 years but ≤ 75 years
* Males or females
* Histological diagnosis of hepatocellular carcinoma
* Curative hepatectomy within the past 4-6 weeks
* ECOG performance status of 0 to 2
* Cardiac functional capacity ≤ to class II (New York Heart Association)
* Patients with adequate renal, hepatic, and haematopoietic function as defined by:

  * Serum creatinine ≤ 2.0 mg/dL
  * Total bilirubin < 2.5 mg/dL
  * Neutrophil count > 1.5 x 10^9/L
  * ALT < 5 x upper limit of normal (ULN)
  * White blood cell (WBC) count ≥ 3 x 10^9/L
  * Platelet count ≥ 80 x 10^9/L
  * Prothrombin time international normalized ratio (PT-INR) ≤ 1.3 (or PT-INR ≤ 1.4 but PT within normal range)
  * Activated partial thromboplastin time (APTT) < ULN

Exclusion Criteria:

* Patients with history of allergy and/or hypersensitivity to anticoagulants/thrombolytic agents, especially heparin.
* Patients with history of immune mediated thrombocytopenia, thrombotic thrombocytopenic purpura, or other platelet disease
* Patients with previous positive result in a heparin-induced thrombocytopenia (HIT) antibody test.
* Patients with any tumour metastasis.
* Patients with uncontrolled infection or serious infection within the past 4 weeks.
* Patients with myocardial infarction, stroke, or congestive heart failure within the past 3 months.
* Patients with history of inflammatory bowel disease, any other abnormal bleeding tendency, or patients at risk of bleeding due to open wounds or planned surgery.
* Patients with acute or chronic gastrointestinal bleeding within the past 1 year.
* Patients with a history of drug abuse or psychiatric disorder.
* Patients with known HIV infection or AIDS-related illness.
* Patients who received other investigational or anti-neoplastic medication within the past 4 weeks.
* Use of aspirin, aspirin-containing medications, non-steroidal anti-inflammatory drugs (except for COX-2 inhibitors), heparin, low molecular weight heparin, warfarin, anti-platelet drugs, or any other anticoagulant medications 2 weeks prior to or during the study period.
* Women who are pregnant or breast-feeding.
* Women of child-bearing potential who are not using an adequate method of contraception.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2004-06; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Jer Chen, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (6):
- Taiwan (6):
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital-Linkou Medical Centre, Taoyuan District

REFERENCES:
- [Derived] Liu CJ, Chang J, Lee PH, Lin DY, Wu CC, Jeng LB, Lin YJ, Mok KT, Lee WC, Yeh HZ, Ho MC, Yang SS, Yang MD, Yu MC, Hu RH, Peng CY, Lai KL, Chang SS, Chen PJ. Adjuvant heparanase inhibitor PI-88 therapy for hepatocellular carcinoma recurrence. World J Gastroenterol. 2014 Aug 28;20(32):11384-93. doi: 10.3748/wjg.v20.i32.11384. PMID 25170226
- [Derived] Liu CJ, Lee PH, Lin DY, Wu CC, Jeng LB, Lin PW, Mok KT, Lee WC, Yeh HZ, Ho MC, Yang SS, Lee CC, Yu MC, Hu RH, Peng CY, Lai KL, Chang SS, Chen PJ. Heparanase inhibitor PI-88 as adjuvant therapy for hepatocellular carcinoma after curative resection: a randomized phase II trial for safety and optimal dosage. J Hepatol. 2009 May;50(5):958-68. doi: 10.1016/j.jhep.2008.12.023. Epub 2009 Feb 15. PMID 19303160

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 215 patients were screened between June 2004 and December 2006. Patients were randomized in balanced blocks per center.
Groups:
- Group A - Untreated Control: untreated control with standard of care
- Group B - 160 mg PI-88/Day: 160 mg PI-88 via subcutaneous injection for four consecutive days per week, every week
- Group C - 250 mg PI-88/Day: 250 mg PI-88 via subcutaneous injection for four consecutive days per week, every week
Period: Overall Study
Arm/Group | Group A - Untreated Control | Group B - 160 mg PI-88/Day | Group C - 250 mg PI-88/Day
Started | 58 | 57 | 57
Completed | 55 | 51 | 43
Not Completed | 3 | 6 | 14

BASELINE CHARACTERISTICS:
Population: ITT population, defined as all randomized subjects who had received at least one dose of study medication (if in a treatment arm) and who had undergone at least one study visit following randomization, including an abdominal CT scan.
Groups:
- Group A - Untreated Control: untreated control with standard of care, ITT population
- Group B - 160 mg PI-88/Day: 160 mg PI-88 via subcutaneous injection for four consecutive days per week, every week, ITT population
- Group C - 250 mg PI-88/Day: 250 mg PI-88 via subcutaneous injection for four consecutive days per week, every week, ITT population
- Total: Total of all reporting groups
Arm/Group | Group A - Untreated Control | Group B - 160 mg PI-88/Day | Group C - 250 mg PI-88/Day | Total
Number analyzed (Participants) | 58 | 56 | 54 | 168
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.96 (12.54) | 51.47 (12.57) | 52.41 (12.03) | 52.39 (12.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 10 | 10 | 35
  Male | 43 | 46 | 44 | 133
Region of Enrollment [Number; unit: participants]
  Taiwan | 58 | 56 | 54 | 168

OUTCOME MEASURES:

1. Primary Outcome: Tumour Non-recurrence Rate
Description: The tumor non-recurrence rate at the end of the 48-week study period
Time Frame: Week 48
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | Group A - Untreated Control | Group B - 160 mg PI-88/Day | Group C - 250 mg PI-88/Day
Number analyzed (Participants) | 58 | 56 | 54
Participants | 32 | 40 | 35
Statistical Analysis 1: Comparison: Group A - Untreated Control vs Group B - 160 mg PI-88/Day; Test type: Non-Inferiority or Equivalence — Sample size is based on the paper 'Two-stage selection and testing design for comparative clinical trials', Thall, PF, Simon, R and Ellenberg, SS. Biometrika (1988),75,(2),303-310; p = 0.072, Chi-squared
Statistical Analysis 2: Comparison: Group A - Untreated Control vs Group C - 250 mg PI-88/Day; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.298, Chi-squared

2. Secondary Outcome: Time to Recurrence
Description: Time to recurrence during the 48-week study period
Time Frame: until confirmed tumour recurrence, or for a maximum of 48 weeks
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Weeks
Groups:
- Group C - 250 mg PI-88/Day: 160 mg PI-88 via subcutaneous injection for four consecutive days per week, every week
Arm/Group | Group A - Untreated Control | Group B - 160 mg PI-88/Day | Group C - 250 mg PI-88/Day
Number analyzed (Participants) | 58 | 56 | 54
Weeks | NA [NA to NA] — The median TTR was unable to be compared among the three study groups because, in all groups, less than 50% of subjects had documented evidence of tumor recurrence by the end of the study. of tumor recurrence. | NA [NA to NA] — The median TTR was unable to be compared among the three study groups because, in all groups, less than 50% of subjects had documented evidence of tumor recurrence by the end of the study. | NA [NA to NA] — The median TTR was unable to be compared among the three study groups because, in all groups, less than 50% of subjects had documented evidence of tumor recurrence by the end of the study.
Statistical Analysis 1: Comparison: Group A - Untreated Control vs Group B - 160 mg PI-88/Day; Test type: Superiority or Other; p = 0.087, Mantel Haenszel; Hazard Ratio (HR) = 0.59
Statistical Analysis 2: Comparison: Group A - Untreated Control vs Group C - 250 mg PI-88/Day; Test type: Superiority or Other; p = 0.653, Mantel Haenszel; Hazard Ratio (HR) = 0.87

3. Secondary Outcome: Survival Rate
Description: Survival rate at the end of the 48-week study period
Time Frame: Week 48
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | Group A - Untreated Control | Group B - 160 mg PI-88/Day | Group C - 250 mg PI-88/Day
Number analyzed (Participants) | 58 | 56 | 54
Participants | 54 | 51 | 51

ADVERSE EVENTS:
Time Frame: During the course of the study (maximum 48 weeks)
Groups:
- Group A - Untreated Control: untreated control with standard of care in safety population defined as all randomized subjects, who had at least one assessment following randomization.
- Group B - 160 mg PI-88/Day: 160 mg PI-88 via subcutaneous injection for four consecutive days per week, every week, safety population (defined as all randomized subjects, who had at least one assessment following randomization)
- Group C - 250 mg PI-88/Day: 250 mg PI-88 via subcutaneous injection for four consecutive days per week, every week, safety population defined as all randomized subjects, who had at least one assessment following randomization
Arm/Group | Group A - Untreated Control | Group B - 160 mg PI-88/Day | Group C - 250 mg PI-88/Day
Serious Adverse Events (participants affected / at risk) | 1/58 | 7/57 | 8/57
Other Adverse Events (participants affected / at risk) | 44/58 | 55/57 | 54/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A - Untreated Control (N=58) | Group B - 160 mg PI-88/Day (N=57) | Group C - 250 mg PI-88/Day (N=57)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Unrelated to treatment
Carbuncle (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Unlikely related to treatment
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) — Unlikely related to treatment
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Unrelated to treatment
Edema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) — Unrelated to treatment
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — Unrelated to treatment
Gastric ulcer hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Unrelated to treatment
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) — Unrelated to treatment (group A); unlikely related to treatment (group B)
Gingival bleeding (General disorders) | 0 (0) | 0 (0) | 1 (1) — Possibly related
Hemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) — Possibly related
Hemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Possibly related
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Unlikely related to treatment
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) — Possibly related
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) — Unlikely related to treatment
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) — Unlikely related to treatment
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) — Unrelated to treatment
Hypovalemic shock (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) — Unlikely related to treatment
Ileus (General disorders) | 0 (0) | 1 (1) | 1 (1) — Unrelated to treatment (group B); unlikely related to treatment (group C)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) — Unlikely related to treatment
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — Unrelated to treatment
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Unlikely related to treatment
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — Unrelated to treatment
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Unrelated to treatment
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — Unrelated to treatment
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Unrelated to treatment
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Unlikely related to treatment
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A - Untreated Control (N=58) | Group B - 160 mg PI-88/Day (N=57) | Group C - 250 mg PI-88/Day (N=57)
ALT increased (Investigations) | 4 (6) | 14 (21) | 19 (33)
APPT prolonged (Investigations) | 0 (0) | 20 (20) | 18 (22)
AST increased (Investigations) | 3 (3) | 10 (18) | 13 (24)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 8 (8) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 5 (5) | 6 (6) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 6 (6) | 5 (6)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 5 (7) | 8 (8)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (7) | 13 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 1 (2)
Ascites (Gastrointestinal disorders) | 1 (1) | 6 (9) | 4 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 5 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (8) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 7 (9) | 3 (3)
Dizziness (Nervous system disorders) | 5 (6) | 1 (2) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 1 (1)
Fatigue (General disorders) | 1 (1) | 3 (3) | 3 (6)
Headache (Nervous system disorders) | 2 (3) | 3 (3) | 4 (4)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 3 (4)
Hyperalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (5) | 1 (1)
Injection site haemorrhage (General disorders) | 0 (0) | 7 (8) | 9 (9)
Injection site pain (General disorders) | 0 (0) | 6 (6) | 4 (4)
Injection site reaction (General disorders) | 0 (0) | 4 (6) | 4 (4)
Insomnia (Psychiatric disorders) | 10 (10) | 11 (13) | 11 (16)
Malaise (General disorders) | 3 (3) | 4 (5) | 5 (6)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 3 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (2) | 1 (3) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 5 (5)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 3 (3) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 6 (20) | 4 (24)
Oedema peripheral (General disorders) | 1 (1) | 4 (4) | 4 (7)
PT prolongation (Investigations) | 0 (0) | 0 (0) | 3 (3)
Periodontits (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5) | 1 (1)
Puritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 3 (3)
Sleep disorders (Psychiatric disorders) | 1 (1) | 1 (1) | 3 (3)
Splenomegaly (Blood and lymphatic system disorders) | 3 (3) | 7 (7) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 6 (14) | 7 (18)
Upper respiratory tract infection (Infections and infestations) | 14 (15) | 8 (8) | 10 (12)
Wound complication (Injury, poisoning and procedural complications) | 2 (3) | 5 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No